CLINICAL TRIAL: NCT00964470
Title: Multi-Center, Prospective, Randomized, Comparison of AWBAT™-D vs. Xeroform™ or Glucan II™ for Treatment of Donor Sites in Burn Surgery
Acronym: AWBAT-D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aubrey Inc. (Industry)
Responsible Party: Stephen Moss/President, Aubrey Inc.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #AW-101008MC-DS
Record Dates: First submitted 2009-08-23; First posted 2009-08-25 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2009-09

CONDITIONS: Treatment of Donor Site Burns
Keywords: Burn, donor site, skin graft, dressing, AWBAT™-D, XEROFORM™, GLUCAN II™
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: AWBAT™-D and XEROFORM™ OR GLUCAN II™ dressings — Dressing, donor site dressings
  Other Names: AWBAT™-D and XEROFORM™ OR GLUCAN II™ donor site dressings

SUMMARY:
The purpose of this study is to compare the rate of healing and the non-adherence of three types of dressings. The study will also compare rate of infection, scarring and perception of pain associated with treatment.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate AWBAT™-D compared to Xeroform™ or Glucan II™ for the treatment of donor sites in burn surgery.

Primary Study Goals:

* To compare the rate of healing of donor sites.
* To compare patient reported perception of pain
* To compare the potential clinical complication rates of:

  * non-adherence,
  * seroma
  * hematoma
  * infection

Secondary Study Goal:

• To compare clinical outcome of donor sites: scarring based on the Vancouver Scar Scale.

ELIGIBILITY:
Inclusion Criteria:

* Burn wounds measuring 1% - 30% TBSA requiring skin grafting
* Anterior bilateral donor sites of approximately the same size taken from the thighs or abdomen

Exclusion Criteria:

* Ventilator dependence
* Pregnancy /Lactation
* Mechanism of injury was electrical, chemical or frostbite
* Co-morbidity which may compromise healing
* Known allergy to porcine or porcine products

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
• To compare the rate of healing of donor sites. • To compare patient reported perception of pain • To compare the potential clinical complication rates of: o non-adherence, o seroma o hematoma o infection | 2 year follow-up

SECONDARY OUTCOMES:
• To compare clinical outcome of donor sites: scarring based on the Vancouver Scar Scale. | 2 year follow-up

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Wishard Health Services Burn Center, Indianapolis, Indiana
  - The University Hospital Burn Center Cincinnati, Cincinnati, Ohio
  - Firefighter's Regional Burn Center, Memphis, Tennessee